CLINICAL TRIAL: NCT04079283
Title: Radiomics of Immunotherapeutics Response Evaluation and Prediction in Solid Tumor: A Multicenter Diagnostic Study
Brief Title: Radiomics of Immunotherapeutics Response Evaluation and Prediction
Acronym: RIREP
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Tianjin Chest Hospital (Other); Shandong Tumor Hospital (Other); West China Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Sun Yat-sen University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Liaoning Cancer Hospital & Institute (Other); Hubei Cancer Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT0100
Record Dates: First submitted 2019-09-01; First posted 2019-09-06 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumor; Predictive Cancer Model
Keywords: Response Evaluation Criteria in Solid Tumors; Computed Tomography; Radiomics; Immunotherapy
MeSH Terms: interventions — Latent Class Analysis; Postmortem Imaging; Radiomics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Monotherapy: Patients who has received mono-therapy of immune checkpoint inhibitor.
  Interventions: Diagnostic Test: Clinical; Diagnostic Test: Semantic; Diagnostic Test: Radiomic
- Combined therapy: Patients who has received immune checkpoint inhibitor combining chemotherapy.
  Interventions: Diagnostic Test: Clinical; Diagnostic Test: Semantic; Diagnostic Test: Radiomic

INTERVENTIONS:
Diagnostic Test: Clinical — Clinical: A diagnostic model incorporating clinical variables (Age, Pathological diagnosis, level of serum tumor biomarkers etc.)
Diagnostic Test: Semantic — Semantic: A diagnostic model incorporating semantic radiological features (shape, location, border, density etc.)
  Other Names: Radiological
Diagnostic Test: Radiomic — Radiomic: A diagnostic model incorporating quantitative radiomic features (histogram, texture, morphology etc.)

SUMMARY:
This study aims to investigate the feasibility and efficiency of CT radiomic analysis which serves as a high through-put analytical strategy applied to image big-data resource in evaluating and predicting the response of immunotherapeutics. A multi-center retrospective diagnostic test has been designed for this aim to compare the predictive performance of clinical model, qualitative model incorporating semantic CT features and image-based quantitative radiomic model. The reference standard of therapeutic effect is determined by the latest evaluation result utilizing iRECIST within 365 days after recruited. This study intends to enroll 400 participates who had been diagnosed with advanced somatic solid tumor confirmed by histo- or cyto-pathological examination and were planning to receive immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathological or cytopathological confirmed solid tumor (including metastatic solid tumor).
2. Patients ≥ 18 years of age on the day of baseline CT scan.
3. Patients received immune checkpoint inhibitors (ICI) monotherapy or combined with chemotherapy in any line of treatment.
4. Patients with at least one measurable target lesion of which minor axis was greater than 15mm and without any local treatment.
5. Female with a negative pregnancy test, or male who agree to use barrier methods of contraception through the therapy period.
6. Patients with a Eastern Cooperative Oncology Group(ECOG) performance status score of 0 or 1.
7. Patients underwent follow-up CT scans with an 6-9-week interval until 365 days after baseline CT scan.
8. Patients with baseline and follow-up CT scans which meet the following conditions: a) Spiral computed tomography device of General Electric Healthcare or Siemens with greater than 16 rows of detectors ; b) Peak kilovoltage: 120kV; c) Dose: auto or fixed; d) Slice resolution: not less than 512 pixels multiply 512 pixels; e) Scanning range: from supraclavicular region to 2cm below the costophrenic angle for thorax, and from diaphragm to pubic symphysis for abdomen; f) contrast-enhanced scan utilizing nonionic low- or iso-osmolar contrast agent and including arterial phase, venous phase and delayed phase at least.

Exclusion Criteria:

1. Patients received any kinds of cytotoxic drugs or experimental drugs 2 weeks before enrollment.
2. Patients meet the contraindications of contrast-enhanced CT scan.
3. Patients who were not suitable for continuous follow-up CT scans.
4. Patients with severe myocardial infarction confirmed by ECG or left ventricular ejection fraction(LVEF) less than 40% or glomerular filtration rate(GFR) less than 45ml/min.
5. Patients who cannot tolerate immunotherapy or with serious immune-related adverse response.
6. Patients with severe interstitial pneumonia confirmed by baseline CT scan.
7. Patients who cannot complete follow-up examinations scheduled by study design.
8. Patients with AIDS or positive serum HIV antibodies.
9. Patients with a CT scan presenting extremely low signal noise ratio or too much artifacts at any timepoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient records in each involved research center from 2017.01.01 to 2019.12.31.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Area Under the receiver operating characteristic curve (ROC) | 6 months and 1 year since course start (365 days)
  Area under curve (AUC) of each diagnostic model

SECONDARY OUTCOMES:
Disease Control Rate | 6 months and 1 year since course start (365 days)
  Disease Control Rate of immunotherapy
Incidence | Through study completion, an average of 1 year
  Incidence of immune-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Ye, M.D, Ph.D, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute And Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided